CLINICAL TRIAL: NCT06797921
Title: Analysis of the Hospital Node in the Management of Acute Events of Patients Referred to Pediatric Palliative Care
Acronym: NO_SCUSE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: NOsCUsE
Record Dates: First submitted 2024-12-03; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Palliative Care
Keywords: pediatric palliative care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to analyze the role of the hospital node in the acute event management of pediatric patients referred to Pediatric Palliative Care. Patients eligible for pediatric palliative care experience frequent hospitalizations. In oncology patients, hospitalizations are mainly for the treatment of the disease and the performance of diagnostic and/or therapeutic procedures, whereas in the case of non-oncology children, admissions occur particularly for the occurrence of complications, which may affect different organs and systems. Hospitalization times are on average longer, so much so that in some cases they can even exceed 100 consecutive days, and have a high risk of re-hospitalization.

DETAILED DESCRIPTION:
In Italy, the prevalence of children needing CPP is estimated at 34-54 per 100,000 population, for a total number between 20,000 and 35,000 children. Prevalence data and projections performed on the British population show that children with life-limiting conditions are progressively increasing. The reason for this increase can be attributed to medical and technological advances that have enabled reductions in neonatal and pediatric mortality and increased the survival of pediatric patients with severe and life-threatening disease. Caring for these patients is complex as they require specific medical and management knowledge and coordination within the health care system. The care of children with medical complexity is interdisciplinary, with different professionals playing a central role for these children. Teamwork is necessary not only for responding to clinical problems but also for defining goals of care and for communication to the patient and family.

ELIGIBILITY:
Inclusion Criteria:

* Living patients aged <18 years at the time of the event
* Patients with conditions eligible for PPCs according to Association for Children's Palliative Care/Royal College of Pediatrics and Child Health

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted with a diagnosis for CPP-candidate diseases at the OUs involved in the study
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of the number of emergency room admissions | through study completion, an average of 1 year
  Number of admissions to the PS
hospital admissions of the pediatric population eligible for Pediatric Palliative Care at the OUs involved in the study. | through study completion, an average of 1 year
  number and duration of hospitalization episodes by year, with prevalence calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Zama, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (7):
- Italy (7):
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Cardiologia Pediatrica, Bologna, Bologna
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Neonatologia e Terapia Intensiva Neonatale, Bologna, Bologna
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Oncoematologia Pediatrica, Bologna, Bologna
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Pediatria d'Urgenza, Pronto Soccorso e Osservazione Breve ed Intensiva, Bologna, Bologna
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Pediatria, Bologna, Bologna
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Rianimazione Pediatrica, Bologna, Bologna
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, U.O.C. Neuropsichiatria dell'età pediatria, Bologna, Bologna

IPD SHARING:
Plan to Share IPD: No